CLINICAL TRIAL: NCT00047502
Title: Phase I Study of Lonafarnib (SCH66336) and Gleevec (Imatinib Mesylate) in Chronic Myelogenous Leukemia (CML)
Brief Title: Study of Lonafarnib and Gleevec in Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID02-221
Record Dates: First submitted 2002-10-08; First posted 2002-10-09 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Chronic Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — lonafarnib; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gleevec + SCH 66336 (Experimental): Participants in CHRONIC PHASE receive Gleevec 400 mg by mouth every day, and SCH66336 100 mg by mouth twice a day.
  Participants in ACCELERATED OR BLASTIC PHASE receive Gleevec 600 mg by mouth every day, and SCH66336 100 mg by mouth twice a day.
  Interventions: Drug: Lonafarnib (SCH66336); Drug: Imatinib Mesylate (Gleevec)

INTERVENTIONS:
Drug: Lonafarnib (SCH66336) — Participants in CHRONIC PHASE receive Gleevec 400 mg by mouth every day, and SCH66336 100 mg by mouth twice a day.
  Participants in ACCELERATED OR BLASTIC PHASE receive SCH66336 100 mg by mouth twice a day.
  Participants in ACCELERATED OR BLASTIC PHASE receive SCH66336 100 mg by mouth twice a day.
  Other Names: SCH66336; Sarasar
Drug: Imatinib Mesylate (Gleevec) — Participants in CHRONIC PHASE receive Gleevec 400 mg by mouth every day.
  Participants in ACCELERATED OR BLASTIC PHASE receive Gleevec 600 mg by mouth every day.
  Other Names: Gleevec; Imatinib; ST1571; NSC-716051

SUMMARY:
The purpose of this study if to investigate the effect of lonafarnib (SCH66336) in combination with Gleevec in the treatment of CML.

DETAILED DESCRIPTION:
Existing pre-clinical and clinical data suggest that SCH66336, a farnesyl transferase inhibitor,exhibits significant activity against CML cells, and in fact may have synergistic activity in combination with imatinib mesylate. Thus, the objectives to the study are (1) to determine the maximum tolerated dose (MTD) and dose limiting toxicities (DLT) of lonafarnib (SCH66336), a farnesyl transferase inhibitor, in combination with imatinib mesylate (Gleevec) in patients with chronic phase, accelerated phase, and blast crisis CML; (2) to assess the pharmacokinetics of the combination of lonafarnib and Gleevec in these patients; and (3) to assess in a preliminary way the biologic activity of the combination of lonafarnib and Gleevec in these patients.

ELIGIBILITY:
1. Patients with Philadelphia chromosome (ph) positive CML in any of the following categories:

   1. Chronic phase patients must have failed therapy with Gleevec. Failure will be defined as: (i) Patients who have not achieved or have lost their hematologic response at 3 months from the start of therapy with Gleevec, or (ii) Patients who have not achieved or have lost their cytogenetic response after 6 months of therapy with Gleevec, or (iii) Patients who have not achieved or have lost their major cytogenetic response after 12 months of therapy with Gleevec.
   2. Patients in accelerated phase, defined as the presence of any of the following features: (i) blasts in peripheral blood (PB) or bone marrow (BM) >/= 15% (but < 30%), (ii) blasts + promyelocytes in PB or BM >/= 30%, (iii) basophils in PB or BM >/= 20%, (iv) platelets < 100 x 10e9/L unrelated to therapy, (v) clonal evolution.
   3. Patients in blast phase, defined by the presence of >/= 30% blasts in peripheral blood and/or bone marrow, or the presence of extramedullary disease.

      2) Patients in accelerated or blastic phase are eligible whether they have received and/or failed Gleevec or not.

      3) Age >/= 16 years.

      4) Patients must sign an informed consent indicating that they are aware of the investigational nature of this study in keeping eith the policies of the hospital. The only acceptable consent form is attached at the end of the protocol.

      5) Performance status </= 2 by Zubrod scale.

      6) Patients must have adequate hepatic functions (bilirubin </= 2.0 mg/dl) and renal functions (creatinine </= 2 mg/dl).

      7) Exclusion criteria:

   <!-- -->

   1. Patients with QTc > 500 msec.
   2. Patients with severe heart disease (cardiac class III and IV) will be excluded.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2002-11-01 (Actual); Primary Completion 2006-04-10 (Actual); Study Completion 2006-04-10 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | 3 months
  Dose-Limiting Toxicity (DLT) defined as grade 3 or 4 non-hematologic toxicity (NCI common criteria, version 2.0). Grade 3 or 4 nausea and vomiting considered DLT only if uncontrolled by antiemetics. Grade 3 or 4 diarrhea considered DLT only if uncontrolled for 48 hours despite adequate antidiarrheal therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge E. Cortes, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org